CLINICAL TRIAL: NCT01198808
Title: Prospective Characterization of Tumor-specific T-cell Immunity in Muscle-invasive Bladder Cancer and Its Correlation With Clinical Parameters
Brief Title: Tumorspecific T-cell Immunity in Bladder Cancer as Prognostic Marker
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: IBT-1
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; chemotherapy; T cells; Immunotherapy; Tumor-specific immunity in bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Bladder cancer is generally susceptible to immunotherapeutic measures. The investigators will characterize 40 patients with muscle-invasive bladder cancer regarding the existence and frequency of tumorspecific T-cells and regulatory T cells. The found data will be correlated to clinical data such as the cancer-specific survival and the response to chemotherapy.

It is hypothesized that those patients with a high number of Tregs and no tumor-specific T-cells have a worse prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed muscle-invasive urothelial carcinoma
* Age > 18 years
* Hemoglobin > 10g/dl
* Signed Informed Consent
* Karnofsky index < 70%

Exclusion Criteria:

* Clinically relevant second malignancy
* Severe comorbidities (e.g. NYHA III, end-stage renal disease)
* Chronic infectious disease (HIV, Tuberculosis)
* Immunosupression
* Severe psychiatric diseases
* Blood donation in the last 4 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with muscle-invasive bladder cancer, who are referred to the university hospital: Krankenhaus rechts der Isar der Technischen Universität München
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Horn, MD, Principal Investigator — Department of Urology, Technische Universität München
Locations (1):
- Urologische Klinik der Technischen Universität München, Munich, Bavaria, Germany